CLINICAL TRIAL: NCT06161012
Title: Evaluation of Delefilcon A and Senofilcon A Daily Disposable Toric Soft Contact Lenses Over Two Weeks of Wear
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CR-6553
Record Dates: First submitted 2023-11-09; First posted 2023-12-07 (Actual); Results first posted 2025-02-26 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Ocular Physiology

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Test/Control (Experimental): Eligible subjects who are habitual soft contact lens wearers will be randomized into the Test/Control sequence, to wear two different study lenses, one at a time, over two wear periods (test then control). Each wear period will be approximately 2 weeks in duration, with a washout period of approximately 1 week between wear periods. Subjects will be advised to wear the study lenses for a minimum of 8 hours per day on at least 5 days per week of each wear period.
  Interventions: Device: Senofilcon A contact lenses (TEST); Device: Delefilcon A contact lenses (CONTROL)
- Control/Test (Experimental): Eligible subjects who are habitual soft contact lens wearers will be randomized into the Control/Test sequence, to wear two different study lenses, one at a time, over two wear periods (control then test). Each wear period will be approximately 2 weeks in duration, with a washout period of approximately 1 week between wear periods. Subjects will be advised to wear the study lenses for a minimum of 8 hours per day on at least 5 days per week of each wear period.
  Interventions: Device: Senofilcon A contact lenses (TEST); Device: Delefilcon A contact lenses (CONTROL)

INTERVENTIONS:
Device: Senofilcon A contact lenses (TEST) — Rotationally stabilized astigmatic soft contact lenses in senofilcon A containing a chromophore to filter High-Energy Visible Light (HEVL)
Device: Delefilcon A contact lenses (CONTROL) — DAILIES TOTAL1® for Astigmatism Contact Lenses (DT1fA)

SUMMARY:
This will be a multi-site, bilateral, dispensing, randomized, controlled, double-masked, 2×2 crossover study to evaluate ocular physiological response.

ELIGIBILITY:
Inclusion Criteria:

Potential subjects must satisfy all of the following criteria to be enrolled in the study.

The subject must:

1. Read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form.
2. Appear able and willing to adhere to the instructions set forth in this clinical protocol.
3. Be between 18 and 39 (inclusive) years of age at the time of screening.
4. By self-report, habitually wear soft contact lenses in both eyes in a daily reusable or daily disposable wear modality (i.e., not extended wear modality). Habitual wear is defined as a minimum of 6 hours of wear per day, for a minimum of 2 days per week during the past four weeks.
5. Possess a wearable pair of spectacles that provide correction for distance vision.
6. In both eyes, have refractive error suitable for correction with the toric contact lens powers available in this study:

   1. Sphere powers (DS) -1.50 through -4.00 in 0.25 steps
   2. Cylinder powers (DC) -0.75 and -1.25
   3. Axes (°) 170, 180, 10, 80, 90, 100
7. Have best corrected monocular distance visual acuity of 20/30 or better in each eye.

Exclusion Criteria:

Potential subjects who meet any of the following criteria will be excluded from participating in the study.

The subject must not:

1. Be currently pregnant or lactating.
2. Be diabetic.
3. Be currently using any ocular medications or have any ocular infection of any type.
4. By self-report, have any ocular or systemic disease, allergies, infection, or use of medication that might contraindicate or interfere with contact lens wear, or otherwise compromise study endpoints, including infectious disease (e.g., hepatitis, tuberculosis), contagious immunosuppressive disease (e.g., Human Immunodeficiency Virus [HIV]), autoimmune disease (e.g., rheumatoid arthritis, Sjögren's syndrome), or history of serious mental illness or seizures. See section 9.1 for additional details regarding excluded systemic medications.
5. Have habitually worn rigid gas permeable (RGP) lenses, orthokeratology lenses, or hybrid lenses (e.g., SynergEyes, SoftPerm) within the past 6 months.
6. Be currently wearing monovision or multifocal contact lenses.
7. Be currently wearing lenses in an extended wear modality.
8. Have a history of strabismus or amblyopia.
9. Be an employee (e.g., Investigator, Coordinator, Technician) or immediate family member of an employee (including partner, child, parent, grandparent, grandchild or sibling of the employee or their spouse) of the clinical site.
10. Have participated in a contact lens or lens care product clinical trial within 7 days prior to study enrollment.
11. Have clinically significant (grade 3 or higher on the FDA grading scale) slit lamp findings (e.g., corneal edema, neovascularization or staining, tarsal abnormalities or bulbar injection) or other corneal or ocular disease or abnormalities that contraindicate contact lens wear or may otherwise compromise study endpoints (including entropion, ectropion, chalazia, recurrent styes, glaucoma, history of recurrent corneal erosions, aphakia, moderate or above corneal distortion, herpetic keratitis).
12. Have fluctuations in vision due to clinically significant dry eye or other ocular conditions.
13. Have had or have planned (within the study period) any ocular or intraocular surgery (e.g., radial keratotomy, PRK, LASIK, iridotomy, retinal laser photocoagulation, etc.).

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 67 (Actual)
Dates: Start 2023-11-16 (Actual); Primary Completion 2024-02-13 (Actual); Study Completion 2024-02-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Vision Care, Inc. Clinical Trial, Study Director — Johnson & Johnson Vision Care, Inc.
Locations (6):
- United States (6):
  - Omega Vision Center, Longwood, Florida
  - Maitland Vision Center - North Orlando Ave, Maitland, Florida
  - ProCare Vision Centers, Granville, Ohio
  - Professional Vision Care Inc. - Westerville, Westerville, Ohio
  - Optometry Group, LLC, Memphis, Tennessee
  - Tyler Eye Associates, Tyler, Texas

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Device Companies have an agreement with the Yale Open Data Access (YODA) to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu
URL: http://yoda.yale.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 67 subjects were enrolled in this study. Of those enrolled, all 67 subjects were dispensed at least one study lens. Of those dispensed, 66 subjects completed the study while one subject was discontinued.
Groups:
- Delefilcon A/ Senofilcon A (C3): Subjects in this sequence were randomized to receive the delefilcon A lens during the first period and the senofilcon A (C3) lens during the second period
- Senofilcon A (C3)\Delefilcon A: Subjects in this sequence were randomized to receive the senofilcon A (C3) lens during the first period and the delefilcon A lens during the second period
Period: Period 1
Arm/Group | Delefilcon A/ Senofilcon A (C3) | Senofilcon A (C3)\Delefilcon A
Started | 33 | 34
Completed | 32 | 34
Not Completed | 1 | 0
Not completed — Unsatisfactory Lens Fitting due to Test Article | 1 | 0
Period: Period 2
Arm/Group | Delefilcon A/ Senofilcon A (C3) | Senofilcon A (C3)\Delefilcon A
Started | 32 | 34
Completed | 32 | 34
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All subjects dispensed at least one study lens.
Groups:
- Total: Subjects dispensed at least one study lens.
Arm/Group | Total
Number analyzed (Participants) | 67
Age, Continuous [Mean (Standard Deviation); unit: Years] | 29.1 (5.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45
  Male | 22
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1
  Black or African American | 3
  White | 61
  Multiple | 2

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Eyes With Grade 3 or Higher Slit Lamp Findings
Description: Slit Lamp Findings (SLF) were assessed using a biomicroscope and was graded using the FDA grading scale (Grade: 0, 1,2, 3 and 4) with grade 0 represents the absence of findings and 1 to 4 representing successively worse findings (i.e. Grade 1 = trace, Grade 2 = Mild, Grade 3 = moderate and Grade 4 = severe). This was performed on each subject eye at every study visit (baseline, unscheduled visits and 1-week follow-up, 2-week follow-up). The data was then dichotomized into two groups. Those with grade 3 or higher and those with grade 2 or lower. The proportion of eyes with SLF with grade 3 or higher was reported for each lens.
Time Frame: Up to 2-Week Follow-up
Population: All dispensed subjects regardless of subsequent withdrawal from study or deviation from protocol.
Measure: Number; unit: Proportion of Eyes
Units Other Than Participants: Eyes
Groups:
- Senofilcon A (C3): Subjects that wore the senofilcon A (C3) lens during either the first or second study periods.
- Delefilcon A: Subjects that wore the delefilcon A lens during either the first or second study periods.
Arm/Group | Senofilcon A (C3) | Delefilcon A
Number analyzed (Participants) | 66 | 66
Number analyzed (Eyes) | 132 | 132
Proportion of Eyes | 0 | 0

ADVERSE EVENTS:
Time Frame: Throughout the entire duration of the study. Approximately five weeks per subject.
Groups:
- Senofilcon A (C3): Subjects that wore the senofilcon A (C3) lens during any of the two study periods.
- Delefilcon A: Subjects that wore the delefilcon A lens during any of the two study periods.
Arm/Group | Senofilcon A (C3) | Delefilcon A
All-Cause Mortality (participants affected / at risk) | 0/66 | 0/67
Serious Adverse Events (participants affected / at risk) | 0/66 | 0/67
Other Adverse Events (participants affected / at risk) | 0/66 | 0/67

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-11-27): https://cdn.clinicaltrials.gov/large-docs/12/NCT06161012/Prot_SAP_000.pdf